CLINICAL TRIAL: NCT02637609
Title: Advancing Stated-preference Methods for Measuring the Preferences of Patients With Type II Diabetes
Brief Title: Measuring the Priorities of Patients With Type II Diabetes Using Likert Scale and Best-worst Scaling
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI 90056532
Record Dates: First submitted 2015-11-18; First posted 2015-12-22 (Estimated); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Type II Diabetes
Keywords: conjoint analysis; stated-preference methods; patient centered outcome research (PCOR); community-based participatory research (CBPR); patient priority; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Likert Scale: Priority elicitation survey using a Likert scale method.
  Interventions: Other: Likert Scale
- Best-Worst Scaling (Case 1): Priority elicitation survey using a best-worst scaling method.
  Interventions: Other: Best-Worst Scaling (Case 1)

INTERVENTIONS:
Other: Likert Scale — Respondents receive questions asking them to rate each barrier or facilitator for diabetes self-management.
  Groups: Likert Scale
Other: Best-Worst Scaling (Case 1) — Respondents receive questions asking them to choose the best and worst factors that affect their diabetes self-management among a list of barriers and facilitators.
  Groups: Best-Worst Scaling (Case 1)

SUMMARY:
In 2012, the FDA Center for Devices and Radiological Health (CDRH) issued guidance to clarify the principal benefit-risk factors FDA considers during the reviews for premarket approval applications and de novo classification requests. In addition to a detailed description of benefits and risks, CDRH listed "patient tolerance for risk and perspective on benefit" as a factor that CDRH may consider in regulatory reviews. It underlined the need for developing methods to measure patient preference and incorporate it into regulatory decision-making. The purpose of this study is to advance methods for patient and community engagement in patient-centered outcome research (PCOR) and has three objectives.

First, demonstrate good practices for patient and community involvement in PCOR projects by applying principles of community-based participatory research (CBPR).

Second, address methodological gaps pertaining to the use of stated-preference methods in studying priorities in PCOR. These include identifying the best methods for identifying patient priorities and strategies for analyzing variation in priorities. The investigators also seek to assess the relevance of stated-preference methods to patients and stakeholders using both qualitative and quantitative methods.

Third, demonstrate good practices for applying stated-preference methods by studying the priorities of patients with type II diabetes. While type II diabetes provides an important case study, this research will advance approaches and methods that will be broadly generalizable to other diseases, and to diverse patient and stakeholder groups.

Clinical Significance:

This project will illustrate and advance methods for assessing the values of patients and stakeholders. It will demonstrate how CBPR methods apply to PCOR studies and the value of stated-preference methods in measuring the priorities of patients and stakeholders and directing health care.

DETAILED DESCRIPTION:
This study will apply the principles of CBPR to involve patients and stakeholders associated with a local community board and a national diabetes advisory board in key decisions in the project. During year 1, the investigators will utilize mixed methods to develop, pretest, and pilot the survey instruments to assess the priorities of patients with type II diabetes. In year 2, the investigators plan further engagement to finalize the survey instruments, and will implement a nationally representative, racially/ethnically diverse sample of patients with type II diabetes. Based on further consultation, the investigators will conduct statistical analysis, including stratified analyses and segmentation of patients with similar priorities. In year 3, mixed methods will be applied to assess beliefs of patients and other consumers about the relevance of this work and its generalizability to other PCOR topics. Finally, lay language reports will be developed to highlight patient and stakeholder engagement and the application of stated-preference methods to the study of the priorities of patients with type II diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participate in the GfK's KnowledgePanel
* Self-reported Type II diabetes diagnosis

Exclusion Criteria:

* Does not have Type II diabetes diagnosis
* Unable to communicate in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type II diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 1103 (Actual)
Dates: Start 2013-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Bridges, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Result] Bridges JFP, Janssen EM, Zhou M, Bone L, Segal JB, Purnell T, Longo DR, Wu A. Comparing Different Ways of Asking People with Type 2 Diabetes about Their Care Priorities and Preferences [Internet]. Washington (DC): Patient-Centered Outcomes Research Institute (PCORI); 2019 May. Available from http://www.ncbi.nlm.nih.gov/books/NBK594947/ PMID 37733885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The survey was conducted through GfK KnowledgePanel. Eligible members were invited by email to participate in the survey. All participants were required to be 18 years or older with self-reported physician-diagnosed type 2 diabetes and able to read English or Spanish. African Americans and Latinos were oversampled.
Pre-assignment Details: 638 respondents (34%) did not respond to the survey and 139 people among those who responded (11%) were excluded based on the screening questions.
Period: Overall Study
Arm/Group | Likert Scale | Best-Worst Scaling (Case 1)
Started | 549 | 554
Completed | 549 | 554
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Respondents who completed the survey.
Groups:
- Likert Scale: Priority measured by Likert scale
  Likert Scale: Respondents receive questions asking them to rate each barrier or facilitator for diabetes self-management.
- Best-Worst Scaling (Case 1): Priority measured by Best-Worse Scaling (BWS)
  Best-Worst Scaling (Case 1): Respondents receive questions asking them to choose the best and worst factors that affect their diabetes self-management among a list of barriers and facilitators.
- Total: Total of all reporting groups
Arm/Group | Likert Scale | Best-Worst Scaling (Case 1) | Total
Number analyzed (Participants) | 549 | 554 | 1103
Age, Continuous [Mean (Full Range); unit: years] | 62.29 [24 to 88] | 61.57 [25 to 91] | 61.93 [24 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 290 | 553
  Male | 286 | 264 | 550
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 287 | 288 | 575
  Black, Non-Hispanic | 126 | 128 | 254
  Other, Non-Hispanic | 12 | 11 | 23
  Hispanic | 117 | 119 | 236
  2+ Races, Non-Hispanic | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 549 | 554 | 1103
Education [Count of Participants; unit: Participants]
  Less than high school | 44 | 38 | 82
  High school | 189 | 173 | 362
  Some college | 163 | 175 | 338
  Bachelor's degree or higher | 153 | 168 | 321
Income [Count of Participants; unit: Participants]
  Less than $25,000 | 132 | 141 | 273
  $25,000 - $49,999 | 156 | 152 | 308
  $50,000 - $74,999 | 106 | 116 | 222
  $75,000 and above | 155 | 145 | 300
Years of diagnosis [Mean (Standard Deviation); unit: years] | 11.54 (8.07) | 11.17 (7.99) | 11.35 (8.03)
Self-reported health [Count of Participants; unit: Participants]
  Excellent | 35 | 25 | 60
  Very good | 170 | 146 | 316
  Good | 227 | 238 | 465
  Fair | 88 | 121 | 209
  Poor | 29 | 24 | 53
No. of hypoglycemic events in the past 6 months [Count of Participants; unit: Participants]
  None | 279 | 292 | 571
  1 time | 80 | 80 | 160
  2-5 times | 147 | 131 | 278
  More than 5 times | 43 | 51 | 94
No. of HbA1c level measured in past 6 months [Count of Participants; unit: Participants]
  None | 30 | 42 | 72
  1 time | 243 | 249 | 492
  More than 2 times | 257 | 250 | 507
  Don't know | 19 | 13 | 32
Most recent HbA1c level [Count of Participants; unit: Participants]
  Over 9.0% | 23 | 35 | 58
  Over 8.0% but under 9.0% | 52 | 53 | 105
  Over 7.0% but under 8.0% | 149 | 148 | 297
  Under 7.0% | 242 | 218 | 460
  Don't know | 83 | 100 | 183
Type of diabetes medicine used [Count of Participants; unit: Participants]
  No prescription medicine | 52 | 47 | 99
  Only pills | 333 | 333 | 666
  Only injections/shots | 48 | 42 | 90
  Pills and injections/shots | 115 | 131 | 246
  Refused | 1 | 1 | 2
Complications [Count of Participants; unit: Participants]
  Yes | 233 | 230 | 463
  No | 316 | 324 | 640
Other chronic conditions [Count of Participants; unit: Participants]
  Yes | 451 | 470 | 921
  No | 98 | 84 | 182

OUTCOME MEASURES:

1. Primary Outcome: Priority Scores for Potential Barriers and Facilitators for Diabetes Self-management
Description: Average Likert score or best-worst score that measures the impact of each factor on diabetes self-management. Positive scores indicate facilitators for diabetes self-management while negative scores indicate barriers. The magnitude of the score suggests the degree of the impact. Both scales are on a +1--1 scale. Positive 1 would be the largest possible facilitator and a negative 1 would be the largest possible barrier.
Time Frame: One-time survey
Population: Respondents who completed the survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Likert Scale: Priority measured by 5-point Likert scale
  Likert Scale: Respondents receive questions asking them to rate each barrier or facilitator for diabetes self-management.
- Best-Worst Scaling (Case 1): Priority measured by best-worst scaling
  Best-Worst Scaling (Case 1): Respondents receive questions asking them to choose the best and worst factors that affect their diabetes self-management among a list of barriers and facilitators.
Arm/Group | Likert Scale | Best-Worst Scaling (Case 1)
Number analyzed (Participants) | 549 | 554
units on a scale
  Healthcare providers | 0.505 [0.433 to 0.577] | 0.327 [0.306 to 0.349]
  My own knowledge | 0.500 [0.437 to 0.563] | 0.369 [0.346 to 0.392]
  Access to healthy food | 0.439 [0.367 to 0.510] | 0.211 [0.187 to 0.235]
  Support from others | 0.359 [0.291 to 0.426] | 0.058 [0.035 to 0.080]
  Staying motivated | 0.344 [0.264 to 0.424] | 0.019 [-0.009 to 0.048]
  Family commitments | 0.293 [0.220 to 0.366] | 0.002 [-0.018 to 0.022]
  Physical environment | 0.287 [0.215 to 0.358] | -0.079 [-0.100 to -0.059]
  My ability to pay | 0.207 [0.119 to 0.295] | -0.166 [-0.189 to -0.143]
  Local events | 0.087 [0.029 to 0.145] | -0.236 [-0.255 to -0.217]
  Work commitments | 0.082 [0.011 to 0.153] | -0.217 [-0.235 to -0.199]
  Other health conditions | 0.067 [-0.013 to 0.147] | -0.281 [-0.303 to -0.259]

2. Secondary Outcome: Self-reported Difficulty in Understanding and Answering the Survey Questions
Description: Questions that asked respondents to evaluate whether it was easy to understand and answer the Likert scale or BWS tasks.
Time Frame: One-time survey
Population: Respondents who completed the survey.
Measure: Count of Participants; unit: Participants
Groups:
- Best-Worst Scaling (Case 1): Priority measured by BWS
  Best-Worst Scaling (Case 1): Respondents receive questions asking them to choose the best and worst factors that affect their diabetes self-management among a list of barriers and facilitators.
Arm/Group | Likert Scale | Best-Worst Scaling (Case 1)
Number analyzed (Participants) | 549 | 554
Participants
  I found it easy to understand the questions: Strongly disagree | 10 | 26
  I found it easy to understand the questions: Disagree | 23 | 90
  I found it easy to understand the questions: Neither agree nor disagree | 73 | 141
  I found it easy to understand the questions: Agree | 316 | 224
  I found it easy to understand the questions: Strongly agree | 122 | 71
  I found it easy to understand the questions: Refused | 5 | 2
  I found it easy to answer all the questions: Strongly disagree | 9 | 34
  I found it easy to answer all the questions: Disagree | 33 | 97
  I found it easy to answer all the questions: Neither agree nor disagree | 71 | 160
  I found it easy to answer all the questions: Agree | 317 | 196
  I found it easy to answer all the questions: Strongly agree | 113 | 66
  I found it easy to answer all the questions: Refused | 6 | 1
  My answers are consistent with my preferences: Strongly disagree | 6 | 6
  My answers are consistent with my preferences: Disagree | 8 | 13
  My answers are consistent with my preferences: Neither agree nor disagree | 61 | 130
  My answers are consistent with my preferences: Agree | 338 | 306
  My answers are consistent with my preferences: Strongly agree | 130 | 99
  My answers are consistent with my preferences: Refused | 6 | 0

ADVERSE EVENTS:
Description: Adverse events not collected
Arm/Group | Likert Scale | Best-Worst Scaling (Case 1)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2014-09-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT02637609/Prot_000.pdf